CLINICAL TRIAL: NCT00989690
Title: Randomized Proteomic Stratified Phase III Study of Second-Line Erlotinib Versus Chemotherapy in Patients With Inoperable Non Small Cell Lung Cancer
Brief Title: Study of Blood and Tissue Samples in Predicting Response to Second-Line Therapy Using Erlotinib Hydrochloride or Chemotherapy in Patients With Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Scientifico H. San Raffaele (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: SRSI-HSRL-02-2007; CDR0000652115 (Registry Identifier: PDQ (Physician Data Query)); 2007-006299-13; EU-20975
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Erlotinib Hydrochloride; Pemetrexed; In Situ Hybridization, Fluorescence; Immunohistochemistry

INTERVENTIONS:
Drug: docetaxel
Drug: erlotinib hydrochloride
Drug: pemetrexed disodium
Genetic: fluorescence in situ hybridization
Genetic: mutation analysis
Genetic: proteomic profiling
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry
Procedure: breath test

SUMMARY:
RATIONALE: Studying the proteins expressed in samples of blood and tissue from patients with cancer may help doctors identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This randomized phase III trial is studying blood and tissue samples in predicting response to second-line therapy using erlotinib hydrochloride or chemotherapy in patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the predictive value of proteomic profiling on the effect of second-line therapy with erlotinib hydrochloride vs standard chemotherapy (pemetrexed disodium or docetaxel) in patients with advanced non-small cell lung cancer.
* To assess the role of other known tissue-based predictive markers (e.g., EGFR-gene copy number, EGFR-protein expression, pAkt, pMAPK, EGFR mutations, EMT markers, and k-Ras mutation).

OUTLINE: This is a multicenter study. Patients are stratified according to smoking status, performance status, proteomic profile, and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive standard chemotherapy with pemetrexed disodium, docetaxel, or another standard drug.
* Arm II: Patients receive standard non-chemotherapy treatment with erlotinib hydrochloride.

Serum is collected after failure of first-line therapy for proteomic analysis by matrix-associated laser desorption/ionization-time of flight. Tissue and blood samples are collected periodically for analysis including EGFR based on IHC and FISH, EGFR and k-Ras mutations, pAkt, pMAPK by IHC, and EMT markers based on IHC and breath condensate protein profile.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC)

  * Advanced NSCLC (stage IIIB or IV)
* Measurable disease
* Underwent previous treatment with 1 non-tyrosine kinase inhibitor as first-line therapy for advanced NSCLC
* No clinical evidence of uncontrolled brain metastases

PATIENT CHARACTERISTICS:

* Caucasian
* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) (≤ 2.5 times ULN in patients with known liver metastases)
* ALT or AST ≤ 3 times ULN (≤ 5 times ULN in patients with known liver metastases)
* Creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Able to comply with planned study procedures
* No multiple severe diseases that can compromise safety (cardiac and renal failure, peripheral neuropathy)
* No other malignancy (except for basal cell skin carcinoma) or pre-neoplastic condition requiring chemotherapeutic treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior surgery or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival
Overall response rate according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Vanesa Gregor, MD, Principal Investigator — Istituto Scientifico H. San Raffaele
Locations (1):
- Istituto Scientifico H. San Raffaele, Milan, Italy

REFERENCES:
- [Derived] Gregorc V, Novello S, Lazzari C, Barni S, Aieta M, Mencoboni M, Grossi F, De Pas T, de Marinis F, Bearz A, Floriani I, Torri V, Bulotta A, Cattaneo A, Grigorieva J, Tsypin M, Roder J, Doglioni C, Levra MG, Petrelli F, Foti S, Vigano M, Bachi A, Roder H. Predictive value of a proteomic signature in patients with non-small-cell lung cancer treated with second-line erlotinib or chemotherapy (PROSE): a biomarker-stratified, randomised phase 3 trial. Lancet Oncol. 2014 Jun;15(7):713-21. doi: 10.1016/S1470-2045(14)70162-7. Epub 2014 May 13. PMID 24831979